CLINICAL TRIAL: NCT03998514
Title: A Phase 1a/1b Study of Safety, Tolerability, and Pharmacokinetics of CB4211 in Healthy Non-obese Subjects and Subjects With Nonalcoholic Fatty Liver Disease
Brief Title: A Phase 1a/1b Study of CB4211 in Healthy Non-obese Subjects and Subjects With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CohBar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CB-4211-001
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Fatty Liver Disease; Liver Disease; Fatty Liver; Nonalcoholic Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver

STUDY DESIGN:
Intervention Model Description: This is a 3-part, randomized, double-blind, placebo-controlled study evaluating the safety, tolerability, PK, and PD of single- and multiple-ascending SC doses of CB4211 in healthy subjects and subjects with NAFLD. Study treatment (CB4211 or placebo) will be administered SC into the abdomen (and if needed, upper and lower thigh) as bolus injections.
Who Masked: Participant, Care Provider, Investigator
Masking Description: randomized, double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Group A1 single ascending dose (SAD) (Experimental): CB4211 Dose 1 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: CB4211 Dose 1; Drug: Placebo
- Group A2 SAD (Experimental): CB4211 Dose 2 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: CB4211 Dose 2; Drug: Placebo
- Group A3 SAD (Experimental): CB4211 Dose 3 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: CB4211 Dose 3; Drug: Placebo
- Group A4 SAD (Experimental): CB4211 Dose 4 (N=1) Placebo (N=1) Subcutaneous injection
  Interventions: Drug: CB4211 Dose 4; Drug: Placebo
- Group A5 SAD (Experimental): CB4211 Dose 5 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: CB4211 Dose 5; Drug: Placebo
- Group A6 SAD (Experimental): CB4211 Dose 6 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: CB4211 Dose 6; Drug: Placebo
- Group B1 multiple ascending dose (MAD) (Experimental): CB4211 Dose to be determined (TBD) (N=6) Placebo (N=2) Subcutaneous injection once daily for 7 days
  Interventions: Drug: CB4211 Dose TBD; Drug: Placebo
- Group B2 MAD (Experimental): CB4211 Dose TBD (N=6) Placebo (N=2) Subcutaneous injection once daily for 7 days
  Interventions: Drug: CB4211 Dose TBD; Drug: Placebo
- Group B3 MAD (Experimental): CB4211 Dose TBD (N=6) Placebo (N=2) Subcutaneous injection once daily for 7 days
  Interventions: Drug: CB4211 Dose TBD; Drug: Placebo
- Part C (Experimental): CB4211 Dose TBD (N=10) Placebo (N=10) Subcutaneous injection once daily for 28 days
  Interventions: Drug: CB4211 Dose TBD; Drug: Placebo

INTERVENTIONS:
Drug: CB4211 Dose 1 — Administered by subcutaneous injection
  Arms: Group A1 single ascending dose (SAD)
Drug: CB4211 Dose 2 — Administered by subcutaneous injection
  Arms: Group A2 SAD
Drug: CB4211 Dose 3 — Administered by subcutaneous injection
  Arms: Group A3 SAD
Drug: CB4211 Dose 4 — Administered by subcutaneous injection
  Arms: Group A4 SAD
Drug: CB4211 Dose 5 — Administered by subcutaneous injection
  Arms: Group A5 SAD
Drug: CB4211 Dose 6 — Administered by subcutaneous injection
  Arms: Group A6 SAD
Drug: CB4211 Dose TBD — Administered by subcutaneous injection
  Arms: Group B1 multiple ascending dose (MAD); Group B2 MAD; Group B3 MAD; Part C
Drug: Placebo — Administered by subcutaneous injection

SUMMARY:
This is a 3 part, randomized, double blind, placebo controlled study evaluating the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple ascending subcutaneous (SC) doses of CB4211 in healthy non obese subjects and subjects with NAFLD.

DETAILED DESCRIPTION:
Part A: Part A is a randomized, double blind, placebo controlled, single ascending dose sequential group study evaluating the safety, tolerability, PK, and PD of a single SC dose of CB4211 in healthy non obese subjects.

Part B: Part B is a randomized, double blind, placebo controlled, multiple ascending dose sequential group study evaluating the safety, tolerability, PK, and PD of once daily SC doses of CB4211 over 7 days in healthy non obese subjects.

Part C: Part C is a randomized, double blind, placebo controlled, multiple dose, parallel group study evaluating the safety, tolerability, PK, and PD of once daily SC doses of CB4211 over 28 days in subjects with NAFLD.

ELIGIBILITY:
Parts A and B Inclusion Criteria:

1. Males or females of nonchildbearing potential, of any race, 18 to 60 years of age, inclusive, at Screening.

   Females of nonchildbearing potential are defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) confirmed by history or postmenopausal (defined as at least 12 continuous months without menses and follicle-stimulating hormone (FSH) ≥40 milli-International unit (mIU)/L and without an alternative medical cause).
2. Body mass index between 18.0 and 30.0 kg/m2 , inclusive, with a minimum body weight of 50.0 kg at Screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening or Check-in as assessed by the Investigator (or designee).
4. Males will agree to use contraception.
5. Has maintained stable weight (by history) for at least 4 weeks prior to Screening.
6. Agrees to the following:

   * Not to initiate a weight-loss program from Screening until the Follow-up visit;
   * To refrain from strenuous exercise from 7 days before Check-in until the Follow-up visit;
   * To maintain consistent dietary habits and exercise routines for the duration of the study.
7. Must have transaminases (aspartate aminotransferase (AST) and alanine aminotransferase (ALT)) and total bilirubin within the normal range at Screening and Check-in. For other laboratory evaluations, the subject may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant.
8. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Parts A and B Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. Clinically significant ECG abnormalities or QT interval corrected for heart rate using Fridericia's method (QTcF) >450 milliseconds for males and >470 milliseconds for females at either Screening or Check-in, or any prior history of QT abnormality.
3. Creatinine clearance of <90 mL/min at Screening, determined using the Cockcroft-Gault (C-G) equation.
4. History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
5. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
6. History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
7. Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
8. Positive urine drug screen (confirmed by repeat) at Screening or positive alcohol breath or urine test result or positive urine drug screen at Check-in.
9. Positive hepatitis panel and/or positive human immunodeficiency virus test. Subjects with serologic finding of immunity consistent with history of prior hepatitis B vaccination may be enrolled.
10. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing or have received a biological product within 3 months or 5 elimination half-lives (whichever is longer) prior to dosing.
11. Use of prescription drugs, nonprescription drugs, dietary supplements including Vitamin E, herbal supplements, hormonal therapy/replacement, or CYP3A4 substrates, inducers and inhibitors within 14 days prior to the first dose of study drug unless, in the opinion of the Investigator and Sponsor's Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety.
12. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
13. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 14 days prior to the first dose of study medication, unless deemed acceptable by the Investigator (or designee).
14. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
15. Receipt of blood products within 2 months prior to Check-in.
16. Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
17. Poor peripheral venous access.
18. Have previously completed or withdrawn from this study or any other study investigating CB4211, and have previously received the investigational product.
19. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Part C Inclusion Criteria:

1. Males or females of nonchildbearing potential, of any race, 18 to 60 years of age, inclusive, at Screening.

   Females of nonchildbearing potential are defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) confirmed by history or postmenopausal (defined as at least 12 continuous months without menses and FSH ≥40 mIU/L and without an alternative medical cause).
2. Body mass index ≥30.0 kg/m2, and body weight ≤115 kg at Screening.
3. History of Fatty Liver Index (FLI) score >60, FLI score >60 at Screening, or documented history of fatty liver with imaging results (eg, standard positive ultrasound or Fibroscan controlled attenuation parameter (CAP) >300 decibels (dB)/m) indicating liver fat >10% within 6 months of Screening. A formal diagnosis of nonalcoholic fatty liver disease (NAFLD) is not required.
4. Liver fat content ≥10% as determined by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) within 14 days prior to Check in. One repeat Baseline MRI-PDFF will be allowed if the first value is below 10%, but greater than or equal to 9.5%. The repeat MRI must be within 14 days of the first MRI, and enrollment must be within 14 days of the repeat MRI. The most current MRI will serve as the baseline. (When available, Fibroscan indicating a CAP >300 dB/m within 6 weeks prior to Check-in may be used as a pre-selection test prior to MRI being performed)
5. No history of common causes of secondary hepatic steatosis such as:

   1. Macrovesicular steatosis: excessive alcohol consumption, hepatitis C (genotype 3), Wilson's disease, lipodystrophy, starvation, parenteral nutrition, abetalipoproteinemia, medications (eg, amiodarone, methotrexate, tamoxifen, corticosteroids, or any drug known to affect hepatic steatosis or insulin resistance)
   2. Microvesicular steatosis: Reye's syndrome, medications (valproate, anti-retroviral medicines), acute fatty liver of pregnancy, HELLP syndrome, inborn errors of metabolism (eg, lecithin-cholesterol acyltransferase deficiency, cholesterol ester storage disease, Wolman disease, lysosomal acid lipase deficiency)
6. Glycosylated hemoglobin A1c <7.0 % at Screening.
7. Fasting blood glucose of ≥100 to <126 mg/dL at Screening.
8. Serum triglyceride level ≤500 mg/dL at Screening
9. Have international normalized ratio (INR) < upper limit of normal (ULN) and platelet count >150,000 at Screening and Check-in. For other abnormalities, the subject may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant.
10. In subjects with ALT, AST, alkaline phosphatase (ALP), or total bilirubin > ULN at Screening, the baseline measurement (BLM) should be determined by 2 separate measurements obtained approximately 4 weeks apart. To be eligible for study entry, the Screening ALT, AST, ALP, and total bilirubin must be < ULN or the following criteria must be met prior to randomization:

    1. ALT ≤3 x ULN for both measurements and the difference between the measurements should be <20% of the lower value;
    2. AST ≤3 x ULN for both measurements and the difference between the measurements should be <20% of the lowest value;
    3. ALP ≤3 x ULN for both measurements and the difference between the measurements should be <20% of the lowest value;
    4. Total bilirubin ≤2 x ULN for both measurements and the difference between the measurements should be <20% of the lowest value.
11. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening or Check-in as assessed by the Investigator (or designee).
12. Males must agree to use contraception.
13. Has maintained stable weight (by history) for at least 4 weeks prior to Screening.
14. Agrees to maintain consistent dietary habits and exercise routines for the duration of the study, including avoiding :

    * initiating any weight-loss program from Screening until the Follow-up visit;
    * strenuous exercise from 7 days before Check-in until the Follow-up visit;
15. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Part C Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic/endocrine (except for type 2 diabetes), allergic, dermatological, hepatic (except for NAFLD), renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, or psychiatric disorder, as determined by the Investigator (or designee).
2. Clinically significant ECG abnormalities or QTcF >450 milliseconds for males and 470 milliseconds for females at Screening, or any prior history of QT abnormality.
3. Currently using any antidiabetic medication (eg, insulin, glucagon-like peptide-1 analogs, agonist therapy) other than a stable regimen of metformin (ie, a fixed dose of metformin for >8 weeks at Screening).
4. Use of fibrates or statins within 6 weeks or beta blocker drugs within 2 weeks prior to Check-in and throughout the duration of the study.
5. Use of Vitamin E, agents associated with changes in liver fat, or agents used for treatment of NAFLD or nonalcoholic steatohepatitis (NASH) within 3 months prior to Screening and throughout the duration of the study.
6. Change in body weight >5% within the 3 months prior to Check-in.
7. History of bariatric surgery and any other gastrointestinal surgery relative to weight loss (eg, Roux-en-Y gastric bypass, laparoscopic adjustable gastric banding, sleeve gastrectomy, duodenal switch with biliopancreatic diversion).
8. Claustrophobia or other contraindication to magnetic resonance imaging.
9. Creatinine clearance of <90 mL/min at Screening, determined using the C-G equation.
10. History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
11. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
12. History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
13. Alcohol consumption of >14 units per week for males and >7 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
14. Positive urine drug screen (confirmed by repeat) at Screening or positive alcohol breath or urine test result or positive urine drug screen at Check-in.
15. Positive hepatitis panel and/or positive human immunodeficiency virus test. Subjects with serologic finding of immunity consistent with history of prior hepatitis B vaccination may be enrolled.
16. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing or have received a biological product within 3 months or 5 elimination half-lives (whichever is longer) prior to dosing.
17. Use of prescription drugs, nonprescription drugs, dietary supplements including peroxisome proliferator-activated receptor-γ agonists, drugs known to affect insulin sensitivity, herbal supplements, hormonal therapy/replacement, or CYP3A4 substrates, inducers, and inhibitors within 14 days or 5 elimination half-lives (whichever is longer) prior to the first dose of study drug and throughout the duration of the study unless, in the opinion of the Investigator and Sponsor's Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety.
18. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
19. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 14 days prior to the first dose of study medication and throughout the duration of the study, unless deemed acceptable by the Investigator (or designee).
20. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in and throughout the duration of the study.
21. Receipt of blood products within 2 months prior to Check-in and throughout the duration of the study.
22. Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
23. Poor peripheral venous access.
24. Have previously completed or withdrawn from this study or any other study investigating CB4211, and have previously received the investigational product.
25. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | up to 8 weeks for Part A; up to 9 weeks for Part B; up to 12 weeks for Part C
  Number of participants with treatment-related adverse events and serious adverse events
Clinical laboratory evaluations | 7 days for Part A; 2 weeks for Part B; 5 weeks for Part C
  Number of participants with clinically significant abnormalities in clinical laboratory values
Vital Signs | 7 days for Part A; 2 weeks for Part B; 5 weeks for Part C
  Number of participants with clinically significant abnormalities in vital signs
12-lead ECG parameters | 7 days for Part A; 2 weeks for Part B; 5 weeks for Part C
  Number of participants with clinically significant abnormalities in 12-lead ECGs
Physical examinations | Time Frame: up to 8 weeks for Part A; up to 9 weeks for Part B; up to 12 weeks for Part C
  Number of participants with clinically significant abnormalities in physical examinations
Injection-site assessments | up to 8 weeks for Part A; up to 9 weeks for Part B; up to 12 weeks for Part C
  Number of participants with treatment-related injection site reactions

SECONDARY OUTCOMES:
Area under the blood/plasma concentration time curve from time zero to infinity of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Area under the blood/plasma concentration time curve from time zero to infinity (AUC0-inf)
Area under the blood/plasma concentration time curve from time zero to the time of the last quantifiable concentration of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Area under the blood/plasma concentration time curve from time zero to the time of the last quantifiable concentration (AUC0-t)
Area under the blood/plasma concentration time curve from time zero to 24 hours postdose of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Area under the blood/plasma concentration time curve from time zero to 24 hours postdose (AUC0-24)
Maximum observed blood/plasma concentration of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Maximum observed blood/plasma concentration (Cmax)
Time of the maximum observed blood/plasma concentration of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Time of the maximum observed blood/plasma concentration (Tmax)
Apparent blood/plasma terminal elimination half life of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Apparent blood/plasma terminal elimination half life (t1/2)
Apparent total blood/plasma clearance of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Apparent total blood/plasma clearance (CL/F)
Apparent volume of distribution of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Apparent volume of distribution(Vz/F)
Amount of CB4211 excreted in urine over the sampling interval | 24 hours for Part A, 7 days for Part B
  Amount of CB4211 excreted in urine over the sampling interval (Aeu)
Percentage of CB4211 excreted in urine | 24 hours for Part A, 7 days for Part B
  Percentage of CB4211 excreted in urine (%fe)
Renal clearance of CB4211 | 24 hours for Part A, 7 days for Part B, 28 days for Part C
  Renal clearance (CLr)
Incidence of antidrug antibodies (ADAs) | Sample at Day -1 and 5 to 7 days postdose for Part A, Day -1, Day 9 prior to discharge and 5 to 7 days post final dose for Part B, and Day -1, Days 14 and 28 predose, and 5 to 7 days post final dose for Part C
  Number of participants with antidrug antibodies (ADAs)

OTHER OUTCOMES:
Change from baseline in body weight | 28 days for Part C only
  Change from baseline in body weight
Change from baseline in liver fat (as determined by magnetic resonance imaging-derived proton density fat fraction [MRI-PDFF]) | 28 days for Part C only
  Change from baseline in liver fat (as determined by magnetic resonance imaging-derived proton density fat fraction [MRI-PDFF])
Proportion of subjects achieving various levels of liver fat reduction at end of treatment | 28 days for Part C
  Proportion of subjects achieving various levels of liver fat reduction at end of treatment
Exploratory biomarkers | Samples pre dose and post dose at 4, 8, 12, and 24 hours for Part A, at 7 days for Part B, and at 7, 14, 21 and 28 days for Part C
  For Parts A, B, and C, exploratory biomarker endpoints include glucose, insulin, triglycerides, non-esterified free fatty acids (NEFA), ALT, adiponectin, and other biomarkers may also be measured in an exploratory fashion. Changes from baseline at 24 hours (Part A), Day 7 (Part B) and Days 7, 14, 21, and 28 (Part C) will be assessed in glucose, insulin; triglycerides, NEFA, ALT, adiponectin, and other biomarkers as required.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - ProScietno, Chula Vista, California
  - Covance Clinical Research Unit Inc., Dallas, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang J, Xu L, Yang L, Liu S, Wang Z. Mitochondrial-Derived Peptide MOTS-c Ameliorates Spared Nerve Injury-Induced Neuropathic Pain in Mice by Inhibiting Microglia Activation and Neuronal Oxidative Damage in the Spinal Cord via the AMPK Pathway. ACS Chem Neurosci. 2023 Jun 21;14(12):2362-2374. doi: 10.1021/acschemneuro.3c00140. Epub 2023 Jun 7. PMID 37285113